CLINICAL TRIAL: NCT01624610
Title: Comparing the Effectiveness of Two Diets to Control the Symptoms of Irritable Bowel Syndrome With Diarrhea (IBS-D): a Randomized, Controlled Trial and Gastrointestinal Microbiome Analysis
Brief Title: Comparing the Effectiveness of 2 Diets for Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shanti Eswaran, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMGI-DIETIBS
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Diarrhea; abdominal pain; diet; nutrition
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Abdominal Pain | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet 1 (Active Comparator): Patients randomized to this arm will receive both written and face-to-face advice about how the components of Diet 1 can be used to control their IBS symptoms.
  Interventions: Other: Dietary intervention
- Diet 2 (Active Comparator): Patients randomized to this arm will receive both written and face-to-face advice about how the components of Diet 2 can be used to control their IBS symptoms.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — After a 14 day screening period, subjects will be randomized to 1 of 2 diets to treat their IBS symptoms. They will receive dietary instruction and are expected to remain on this diet for 4 weeks.

SUMMARY:
The purpose of the study is to find out if the diets often recommended for patients with Irritable Bowel Syndrome with diarrhea (IBS-D) provide adequate relief. The study will compare two diets that are used to treat IBS-D symptoms to see which one is more effective. The study will also measure the effect of these diets on the bowel flora, which are the good bacteria that inhabit the bowels in healthy people.

DETAILED DESCRIPTION:
As irritable bowel syndrome (IBS) symptoms are often refractory to conventional therapies, there has been increasing interest in the role of diet in IBS. Certain foods may exacerbate symptoms of IBS. Thus, restricted diets have recently gained attention for the treatment IBS. The mechanism by which symptoms are improved is unclear, but these diets may improve symptoms by exerting changes on the GI microbiome.

Aims:

Primary Objective:

-Compare the proportion of patients with irritable bowel syndrome (IBS-D) reporting adequate relief on Diet 1 vs Diet 2

Secondary Objectives:

* Assess the effects of these diets in patients with diarrhea-predominant IBS on the gastrointestinal microbiota and blood based biomarkers.
* Compare the efficacy of Diet 1 vs Diet 2 in patients with diarrhea-predominant IBS on pre-specified clinical and quality of life endpoints.

Methods:

This is a prospective randomized control trial of adults meeting the Rome III criteria for irritable bowel syndrome with diarrhea (IBS-D). After a 2 week screening period and randomization, during which the severity of symptoms will be assessed and eligibility determined, patients will be randomized to Diet 1 vs Diet 2 for a period of 4 weeks.

The primary endpoint will be a comparison of the proportion of patients in each group reporting adequate relief of their IBS symptoms. For the secondary clinical outcomes, a responder definition incorporating abdominal pain and stool consistency as proposed by the FDA will be utilized. Key IBS-D symptoms will be assessed daily and adequate relief of IBS-D symptoms will be assessed weekly during the randomization period. We will also determine if a difference can be detected with high probability in the relative abundance and variety of specific bacterial taxa between the two groups before and after the 4 week dietary intervention. In addition, blood samples will be collected before and after randomization to measure relevant biomarkers of immune activation.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome III criteria for IBS as assessed by a gastroenterologist:
* Fulfill the Rome III stool consistency criteria for IBS -D
* Willingness to maintain a stable dosage of IBS medications during the pretreatment baseline period, including tricyclic antidepressants; "rescue" medications permitted (ie Loperamide 2mg up to 4 times per day prn diarrhea)
* Ability to provide written informed consent for study participation
* Capable of independently completing all requirements of the study including returning for required visits
* Documentation of normal colonoscopy with colon biopsies within five years
* Documentation of normal TSH, CBC, electrolyte panel
* Negative evaluation for celiac disease either with normal TTG, EMA, and/or duodenal biopsy.

Exclusion Criteria:

* Unable to understand or provide written informed consent
* Pregnancy
* IBS with constipation or mixed subtype
* Comorbid medical problems that may affect gastrointestinal transit or motility:
* Inflammatory bowel disease
* Extraintestinal disease known to affect the gastrointestinal system (ie, scleroderma, unstable thyroid disease, diabetes mellitus, etc.)
* Severe renal or hepatic disease
* Previous abdominal surgery other than appendectomy, cholecystectomy, and gynecologic/urologic surgery
* Previous treatment with some diets for IBS
* Concurrent medications not permitted including probiotics, antibiotics, and narcotics
* Active participation in another form of dietary therapy
* Patients who have undergone surgery to the GI tract except appendectomy or cholecystectomy if performed more than six months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adequate relief. | 4 weeks
  Compare the proportion of patients with irritable bowel syndrome (IBS-D) reporting adequate relief on Diet 1 v Diet 2.

SECONDARY OUTCOMES:
Composite endpoint | 4 weeks
  Composite endpoint: A responder will report a ≥30% reduction in mean daily abdominal pain score and a decrease in mean daily BSFS value of ≥1 compared to baseline for ≥2 of 4 treatment weeks. The proportion of responders between the 2 groups will be compared.
Abdominal Pain | 4 weeks
  An abdominal pain responder will report a ≥30% reduction in mean daily abdominal pain score compared to baseline for ≥2 of 4 treatment weeks. The proportion of responders between the two groups will be compared. Between group differences in the proportion of patients with a ≥30% reduction in mean daily abdominal pain score compared to baseline at the end of each treatment week will also be assessed.
Stool consistency | 4 weeks
  For stool consistency, a responder will be defined as one who reports a decrease in mean daily BSFS value of 1 or more compared to baseline for ≥2 of 4 treatment weeks. The proportion of responders between the 2 groups will be compared. Between group differences in the proportion of patients with a decrease in BSFS value of ≥1 compared to baseline at the end of each treatment week will also be assessed.
Stool frequency | 4 weeks
  The number of bowel movements will be recorded each day by IVRS. The change from baseline in mean daily stool frequency for each treatment week will be compared for the two groups.
Individual symptoms | 4 weeks
  The change from baseline in daily NRS scores averaged over each treatment week for abdominal discomfort, urgency, bloating, and fatigue will compared between the 2 groups.
Quality of life measures | 4 weeks
  IBS-Quality of Life scores, Hospital Depression Anxiety Scores, Work Productivity and Activity Impairment questionnaire, and Sleep Assessment questionnaires will be compared between groups before and after the dietary intervention.
Stool Microbiome | 4 weeks
  The effect of these 2 diets on the gut microbiome (number and species) in the context of IBS is not known. A change in the microbiota may be a mechanism through which symptom response is mediated.
  We will be measuring the shift in the relative abundance (richness) and variety (diversity) of gut microbial taxa in patients with irritable bowel syndrome (IBS-D) in response to dietary intervention. Stool microbiome would be collected and analyzed using the PhyloChip™ Assay (Second Genome Inc., San Bruno, CA).
Serum Biomarker Panel | 4 weeks
  Recent attempts have been made to identify a serological biomarker profile (Prometheus Therapeutics & Diagnostics, San Diego, CA) which accurately identifies patients with IBS. We intend to perform a biomarker test panel at enrollment in all study subjects to assess whether specific combinations of biomarkers can positively or negatively predict response to either diet.

CONTACTS AND LOCATIONS:
Overall Officials: Shanti L Eswaran, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Derived] Eswaran S, Chey WD, Jackson K, Pillai S, Chey SW, Han-Markey T. A Diet Low in Fermentable Oligo-, Di-, and Monosaccharides and Polyols Improves Quality of Life and Reduces Activity Impairment in Patients With Irritable Bowel Syndrome and Diarrhea. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1890-1899.e3. doi: 10.1016/j.cgh.2017.06.044. Epub 2017 Jun 28. PMID 28668539